CLINICAL TRIAL: NCT06603597
Title: Prospective Evaluation of Outcomes for HER2-positive Breast Cancer (PRO-HER2)
Brief Title: HER2-positive Breast Cancer Registry
Acronym: PRO-HER2
Status: Recruiting | Type: Observational
Sponsor: Priyanka Sharma (Other)
Responsible Party: Sponsor-Investigator, Priyanka Sharma, Professor of Medicine, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 160944
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: HER2 + Breast Cancer
Keywords: breast cancer; registry; HER2+; HER2 positive
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood plasma, serum, buffy layer; fixed tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HER2-positive breast cancer: Patients with stage I-IV HER2-positive breast cancer

SUMMARY:
The goal of this observational study is to better understand links between patient or tumor characteristics and outcomes in HER2-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-IV HER2-positive breast cancer

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage I-IV HER2-positive breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2044-10 (Estimated); Study Completion 2044-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | From diagnosis to 5 years after diagnosis
  For patients with stage I-III HER2-positive breast cancer, percentage of patients who are alive at 5 years after diagnosis.

SECONDARY OUTCOMES:
Pathologic complete response rate | From start of neoadjuvant systemic treatment until approximately 8 months after start of neoadjuvant systemic treatment
  Percentage of patients with stage I-III HER2-positive breast cancer who received neoadjuvant systemic therapy and experienced pathologic complete response.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - KUCC - Indian Creek, Overland Park, Kansas
  - KUCC - Overland Park, Overland Park, Kansas
  - KUCC - Briarcliff, Westwood, Kansas
  - KUCC - Olathe, Westwood, Kansas
  - The University of Kansas Cancer Center, Westwood, Kansas
  - KUCC - Lee's Summit, Lee's Summit, Missouri